CLINICAL TRIAL: NCT02572323
Title: Phase II Trial of Tesamorelin for Cognition in Aging HIV-Infected Persons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Southern California (Other); PalmTree Clinical Research Inc. (Unknown); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ronald Ellis, Professor of Neurosciences, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01AG048650 (NIH)
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate group (Active Comparator): 1.4mg of tesamorelin is injected once a day for 6 months, then no treatment is given for 6 months
  Interventions: Drug: Tesamorelin
- Deferred group (Placebo Comparator): No treatment is given for 6 months, then 1.4mg of tesamorelin is injected once a day for 6 months
  Interventions: Drug: Tesamorelin

INTERVENTIONS:
Drug: Tesamorelin — Tesamorelin is an injectable medication already approved by the U.S. FDA to treat abdominal fat accumulation in HIV
  Other Names: Egrifta

SUMMARY:
The aim of this study is to test whether tesamorelin, in combination with a text-messaging application to help with motivation and adherence, will significantly improve memory and thinking in HIV.

DETAILED DESCRIPTION:
HIV infection can result in memory and thinking difficulties in some people, even those successfully treated with antiretroviral medications. Tesamorelin is an injectable medication already approved by the U.S. FDA to treat abdominal fat accumulation in HIV. Abdominal fat accumulation is linked to memory and thinking difficulties, and previous studies have suggested that tesamorelin also may be beneficial for memory and thinking, but this has not been tested in HIV. The aim of this study is to test whether tesamorelin, in combination with a text-messaging application to help with motivation and adherence, will significantly improve memory and thinking in HIV. We plan to enroll 100 volunteers with HIV infection at 2 sites - the University of California, San Diego and the University of Southern California, University of San Francisco and the satellite site, PalmTree Clinical Research, Inc. Before entry, volunteers will be required to show evidence of abdominal obesity and a minimum level of memory and thinking difficulties on cognitive tests. This is a randomized trial in which each volunteer will have a 60% chance of initially receiving tesamorelin (the immediate group) and a 40% chance of initially receiving no treatment (the deferred group). Subsequently, the deferred group (those who initially received no treatment) will receive tesamorelin for 6 months and those who initially received tesamorelin will receive no treatment for 6 months. Volunteers will be trained in the use of a 2-way text-messaging system that will help the research team to support volunteers' ability to take the study medication as directed. We will measure volunteers' memory and thinking skills before and at the end of treatment. We will collect blood at various points during the study to check for safety of the treatment and to determine its effects on the body. Volunteers will also be asked to have magnetic resonance scans of the head and abdomen to monitor the effects of the study medication on brain chemistry and abdominal fat.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by any FDA licensed clinical test including HIV enzyme/antigen test or chemiluminescence immunoassay (E/CIA) or plasma HIV-1 RNA viral load.
* Antiretroviral therapy: Patient currently receiving a combination antiretroviral therapy (cART) regimen ≥12 weeks with no interruptions longer than 7 days and HIV <500 copies/ml during that time.
* Men or women 40 years of age and older
* Abdominal minimal waist circumference ≥ 95cm for men and ≥94cm for women or minimal waist to hip ratio of ≥ 0.88 for women (each based on an average of three separate measurements)
* Screening neuropsychological Global Deficit Score of ≥ 0.35
* The following laboratory values obtained within 90 days prior to entry by any CLIA certified laboratory.

  * Absolute neutrophil count (ANC) ≥750/mm3
  * Hemoglobin ≥8.0 g/dL
  * Platelet count ≥50,000/mm3
  * HgbA1C ≤8.0%
  * Calculated creatinine clearance of ≥20 mL/min as estimated by the Cockroft-Gault formula
  * Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT) <5 X upper limit of normal (ULN) and alkaline phosphatase <3 X upper limit of normal (ULN) without evidence of active liver disease other than non-alcoholic fatty liver disease (NAFLD) or hepatitis C requiring treatment.
  * Total bilirubin ≤2.5 x ULN (if the participant is receiving atazanavir, a total bilirubin of ≤5 x ULN is acceptable).
* For females of reproductive potential, negative serum or urine pregnancy test within 30 days prior to entry by any test performed by a CLIA certified laboratory or is using a point of care (POC)/ CLIA-waived test.
* Contraception requirements: For females of reproductive potential, she or male partner is willing to use a contraceptive during sexual intercourse.
* Ability and willingness of participant or legal guardian/representative to provide informed consent

Exclusion Criteria:

* Clinical contraindications

  * History of neurocognitive confounding conditions that explain current impairment including but not limited to stroke, head injury, psychotic disorder, active substance use disorder by DSM, or opportunistic CNS infection
  * Hepatitis C virus infection defined as HCV antibody positive requiring treatment and plans for treatment during study therapy
  * Active or relapsing autoimmune disorder that may require immunotherapy during this treatment trial
  * Active malignancy other than basal or squamous skin cancer.
* Breastfeeding or pregnancy
* Excluded medications used within the last 90 days: active or planned use of rhGH, anabolic steroids (other than replacement doses of testosterone), anti-TNFa therapy or other biologic (tocilizumab, Xelijanz, etc.)
* Anticipated need to start new daily anti-inflammatory therapy such as NSAIDs (excluding aspirin for vascular prophylaxis), systemic corticosteroids, or anti-malarials, or plan to discontinue regular dosing with these drugs during study treatment.
* Known allergy/sensitivity or any hypersensitivity to tesamorelin
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Acute or serious illness requiring systemic treatment and/or hospitalization within 60 days prior to entry
* Use of tesamorelin in the last 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Neurocognitive performance | 6 months and 12 months
  Change in neurocognitive performance measured by Global Deficit Score (GDS)

SECONDARY OUTCOMES:
Biomarkers of visceral adipose tissue (VAT)-related inflammation and immune activation, metabolic parameters, and neuronal integrity | 6 months
  Change in IGF-1, magnetic resonance spectroscopy measures of brain inflammation/immune activation and hippocampal volume

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Ellis, MD, PhD, Principal Investigator — University of California, San Diego; Fred Sattler, MD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - Keck School of Medicine of the University of Southern California, Los Angeles, California
  - PalmTree, Palm Springs, California
  - HIV Neurobehavioral Research Program (HNRP), San Diego, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No